CLINICAL TRIAL: NCT06469138
Title: A Phase 1, Open-label, Nonrandomized Study to Investigate the Mass Balance Recovery and Metabolic Profile of 14C-bemcentinib Following Single Oral Administration in Healthy Male Subjects
Brief Title: A Study to Investigate 14C-bemcentinib in Healthy Male Subjects
Acronym: 8479217
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BerGenBio ASA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGBC021
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Non-Small Cell Lung Cancer; Metastatic Melanoma; Acute Myeloid Leukemia; Myelodysplastic Syndromes; Metastatic Pancreatic Cancer; Glioblastoma; Malignant Mesothelioma; COVID-19
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Pancreatic Neoplasms; Glioblastoma; Mesothelioma, Malignant; COVID-19 | interventions — bemcentinib

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to active treatment and will be dosed within a single cohort of up to 8 participants (with 6 required to complete).
Masking Description: N/A - study is open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Dose Cohort - 200 mg containing approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib (Experimental): This is the only treatment arm in this study. Up to 8 participants will receive a single oral dose of 200 mg containing approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib, 30 minutes after starting a standard high-fat breakfast.
  Interventions: Drug: Bemcentinib

INTERVENTIONS:
Drug: Bemcentinib — Each 200 mg dose contains approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib and is administered as a single dose on Day 1 of the study.
  Other Names: BGB324

SUMMARY:
The aims of this Study were to determine:

* How much of the Study Drug (bemcentinib) ends up in urine and faeces
* How much of the Study Drug and its breakdown products get into the bloodstream
* The breakdown products (metabolites) of the Study Drug
* The safety of the Study Drug and any side effects that might be associated with it.

DETAILED DESCRIPTION:
This was a Phase 1, open-label, nonrandomized, single oral dose study in up to 8 healthy male subjects (with 6 required to complete the study).

Potential subjects were screened to assess their eligibility to enter the study within 28 days prior to dose administration. Up to 8 subjects were enrolled to ensure that 6 subjects completed the study. Subjects were admitted into the study site on Day -1. On the morning of Day 1, all subjects received a single oral dose of 200 mg containing approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib, 30 minutes after starting a standard high-fat breakfast.

Subjects were confined to the study site until at least Day 8. Subjects were discharged from the study site on Day 8 if the following discharge criteria were met:

·≥90% mass balance recovery, and

·<1% of the total radioactive dose is recovered in combined excreta (urine and feces)in 2 consecutive 24-hour periods.

If these discharge criteria were not met by Day 8, subjects were required to remain resident until discharge criteria are met, up to Day 15. If criteria were not met by Day 15, subjects were asked to collect 24-hour excreta samples on up to 2 further occasions on a nonresidential basis to allow extrapolation of urinary and fecal excretion. If needed, the 2 additional 24-hour nonresidential collections started on the morning of Days 22 and 29 (to be brought into the study site at the end of the collection interval on Days 23 and 30, respectively). If on the second occasion the subject still did not meet the desired criterion, then the subject was discharged from the study, per investigator and sponsor decision.

Subjects experiencing emesis during the first 4 hours post-dose were discharged on the same day from the study site, provided there were no safety concerns, and after discharge study procedures were performed.

The total duration of study participation for each subject (from screening to outpatient visit [if required]) was anticipated to be a maximum of approximately 58 days.

ELIGIBILITY:
Inclusion Criteria:

1. Males of any race, between 35 and 55 years of age, inclusive.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive, and a total body weight between 50 and 100 kg, inclusive.
3. In good health, determined by no clinically significant findings from medical history, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in and from the physical examination at check-in, as assessed by the investigator (or designee).
4. No clinically significant abnormalities in 12-lead ECG determined within 28 days before dose of IMP including average PR > 220 ms and QT interval corrected for heart rate using Fridericia's formula >450 ms.
5. No history of clinically significant dysrhythmias (long QT features on ECG, sustained bradycardia, left bundle branch block, or ventricular arrhythmia), atrial fibrillation, or history of familial long QT syndromes.
6. Will agree to use contraception as detailed in the study protocol.
7. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
8. History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

Medical conditions

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
4. Positive hepatitis panel and/or positive human immunodeficiency virus test.

   Prior/concomitant therapy
5. Administration of a COVID-19 vaccine in the past 30 days prior to dosing.
6. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to check-in, unless deemed acceptable by the investigator (or designee).
7. Use or intend to use any prescription medications/products within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee).
8. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee).
9. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to check-in, unless deemed acceptable by the investigator (or designee).

   Prior/concurrent clinical study experience
10. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to dosing.
11. Subjects who have participated in any clinical study involving a radiolabelled investigational product within 12 months prior to check-in.
12. Have previously completed or withdrawn from this study or any other study investigating bemcentinib, and have previously received bemcentinib.

    Diet and lifestyle
13. Alcohol consumption of > 28 units per week for males. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
14. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at screening or check-in.
15. History of alcoholism or drug/chemical abuse within 2 years prior to check-in.
16. Use of tobacco- or nicotine-containing products within 3 months prior to check-in, or positive cotinine at screening or check-in.
17. Ingestion of poppy seed-, Seville orange-, or grapefruit-containing foods or beverages within 7 days prior to check-in.

    Other exclusions
18. Receipt of blood products within 2 months prior to check-in.
19. Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
20. Poor peripheral venous access.
21. Subjects with exposure to significant diagnostic or therapeutic radiation (eg, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
22. Subjects who, in the opinion of the investigator (or designee), should not participate in this study.

Subjects may previously have been screened on a generic basis to determine their eligibility for inclusion in Phase 1 clinical studies conducted at the study site. If generic screening was performed within the specified study screening window, selected study-specific procedures will be repeated either at an additional screening visit or on admission to the study site on Day -1.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — As this study involves radiation exposures, as per the applicable regulatory guidance, the most relevant population for this study is healthy male volunteers.
Enrollment: 6 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Brooks, MBChB, Principal Investigator — Labcorp Clinical Research Unit Ltd.
Locations (1):
- Labcorp Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No
At this stage, it is not planned that any IPD information will be shared with other researchers outside of the Sponsor and Clinical Research Organisation undertaking the conduct of this study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment was undertaken in the United Kingdom at a single site. The recruitment process began in August 2022 and concluded in September 2022. A sufficient number of volunteers were screened in order to successfully recruit 6 eligible participants.
Pre-assignment Details: Participants were screened to the inclusion/exclusion criteria of the protocol. The following assessments were performed: Informed Consent, Demographics, Medical History, Height & Weight, ECG, Vital Signs and Safety Laboratory Testing/Urinalysis & Drugs of Abuse testing.
Groups:
- Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib: This was the only treatment arm in the study. Up to 8 participants were to receive a single oral dose of 200 mg containing approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib, 30 minutes after starting a standard high-fat breakfast.
  Bemcentinib: Each 200 mg dose contained approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib and was administered as a single dose on Day 1 of the study.
Period: Overall Study
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This analysis population denotes all of the participants enrolled within the baseline analysis i.e., all eligible participants enrolled onto the study who subsequently fully completed.
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (4.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6
Height [Mean (Standard Deviation); unit: Centimetres] | 172.30 (6.508)
Weight [Mean (Standard Deviation); unit: Kilograms] | 80.58 (7.066)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.15 (1.952)

OUTCOME MEASURES:

1. Primary Outcome: Total Radioactivity - Plasma Maximum Observed Concentration (Cmax)
Description: This endpoint will report the relevant data for the parameters assessed in order to measure total radioactivity in plasma (based upon plasma samples collected at set timepoints during the study). Analysis was derived from obtaining plasma samples from participants at set timepoints described and deriving PK parameters through the use of noncompartmental procedures in validated software (WinNonlin Version 8.3.5).
Time Frame: Samples collected over a 2-week period: Days 1-8: Predose, 15 and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours post-dose, Days 8-15: 192, 216, 240, 264, 288, 312, and 336 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
ngEq/mL | 81.2 (26.8)

2. Primary Outcome: Total Radioactivity - Whole Blood Maximum Observed Concentration (Cmax)
Description: This endpoint will report the relevant data for the parameters assessed in order to measure total radioactivity in whole blood (based upon whole blood samples collected at set timepoints during the study). Analysis was derived from obtaining whole blood samples from participants at set timepoints described and deriving PK parameters through the use of noncompartmental procedures in validated software (WinNonlin Version 8.3.5).
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
ngEq/mL | 121 (21.6)

3. Primary Outcome: Plasma Pharmacokinetic Parameters Bemcentinib - Maximum Observed Concentration (Cmax)
Description: Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for 14C-bemcentinib. This endpoint will report the summary of derived pharmacokinetic parameters for the maximum observed concentration (Cmax) of 14C-bemcentinib in plasma. Analysis was derived from obtaining plasma samples from participants at set timepoints described and deriving PK parameters through the use of noncompartmental procedures in validated software (WinNonlin Version 8.3.5).
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
ng/mL | 55.8 (23.5)

4. Primary Outcome: Plasma Pharmacokinetic Parameters Bemcentinib - Time to Maximum Observed Concentration (Tmax)
Description: Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for 14C-bemcentinib. This endpoint will report the summary of derived pharmacokinetic parameters for the time to maximum observed concentration (Tmax) of 14C-bemcentinib in plasma. Analysis was derived from obtaining plasma samples from participants at set timepoints described and deriving PK parameters through the use of noncompartmental procedures in validated software (WinNonlin Version 8.3.5).
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
Hour | 12.0 [12.0 to 36.0]

5. Primary Outcome: Plasma Pharmacokinetic Parameters Bemcentinib - Terminal Elimination Half-life (t1/2)
Description: Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for 14C-bemcentinib. This endpoint will report the summary of derived pharmacokinetic parameters for the terminal elimination half-life (t1/2) of 14C-bemcentinib in plasma. Analysis was derived from obtaining plasma samples from participants at set timepoints described and deriving PK parameters through the use of noncompartmental procedures in validated software (WinNonlin Version 8.3.5).
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
Hour | 92.0 (5.3)

6. Primary Outcome: Plasma Pharmacokinetic Parameters Bemcentinib - Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞)
Description: Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for 14C-bemcentinib. This endpoint will report the summary of derived pharmacokinetic parameters for the area under the concentration-time curve from time 0 extrapolated to infinity (AUC0-∞) of 14C-bemcentinib in plasma. Analysis was derived from obtaining plasma samples from participants at set timepoints described and deriving PK parameters through the use of noncompartmental procedures in validated software (WinNonlin Version 8.3.5).
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
h*ng/mL | 6050 (12.3)

7. Primary Outcome: Plasma Pharmacokinetic Parameters Bemcentinib - Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-tlast)
Description: Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for 14C-bemcentinib. This endpoint will report the summary of derived pharmacokinetic parameters for the area under the concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-tlast) of 14C-bemcentinib in plasma. Analysis was derived from obtaining plasma samples from participants at set timepoints described and deriving PK parameters through the use of noncompartmental procedures in validated software (WinNonlin Version 8.3.5).
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
h*ng/mL | 5550 (13.3)

8. Secondary Outcome: Number of Participants With Adverse Events
Description: This secondary endpoint relates to the number of participants who report an adverse event (AE) during the study.
Time Frame: Collection of AEs occurs through ad hoc reporting from the participants from the point of signature of informed consent through to study completion (up to 5 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
Participants | 3

9. Secondary Outcome: Number of Participants Who Report a Change From Normal Range Values for Laboratory Safety Parameters (Serum Biochemistry, Serum Haematology or Urinalysis) From First Dose on Day 1 to Study Completion.
Description: This secondary endpoint will report the number of participants who record a value which is deemed as outside of the normal range (clinically significant values only) for any of the serum biochemistry, serum haematology or urinalysis parameters as defined in the study protocol following first dose administration on Day 1 up to completion of the study.
Time Frame: From Day 1 to study completion (up to 5 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
Participants | 0

10. Secondary Outcome: Number of Participants Who Report a Change From Normal Range Values for Any of the Associated 12-Lead ECG Parameters From First Dose on Day 1 to Study Completion.
Description: This secondary endpoint will report the number of participants who record a value which is deemed as outside of the normal range (clinically significant values only) for any of the 12-Lead ECG parameters as defined in the study protocol following first dose administration on Day 1 up to completion of the study.
Time Frame: From Day 1 to study completion (up to 5 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
Participants | 0

11. Secondary Outcome: Number of Participants Who Report a Change From Normal Range Values for Any of the Vital Signs Parameters From First Dose on Day 1 to Study Completion.
Description: This secondary endpoint will report the number of participants who record a value which is deemed as outside of the normal range (clinically significant values only) for any of the vital signs parameters as defined in the study protocol following first dose administration on Day 1 up to completion of the study.
Time Frame: From Day 1 to study completion (up to 5 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
Participants | 0

12. Secondary Outcome: Number of Participants Who Report a Change From Normal With Respect to Physical Examination Parameters From First Dose on Day 1 to Study Completion.
Description: This secondary endpoint will report the number of participants who record a change which is deemed as outside of normal range (clinically significant changes only) for any of the physical examination parameters as defined in the study protocol following first dose administration on Day 1 up to completion of the study.
Time Frame: From Day 1 to study completion (up to 5 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported through ad hoc reporting from the participants from the point of signature of informed consent through to study completion (up to 5 weeks).
Arm/Group | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose Cohort - 200 mg Containing Approximately 32.8 μCi (1.21 MBq) of 14C-bemcentinib (N=6)
Headache (Nervous system disorders) | 1 (2) — Headache
Bruising Right Antecubital Fossa (Venepuncture Related) (General disorders) | 1 (1) — Vessel Puncture Site Bruise
Loose Stool (Gastrointestinal disorders) | 1 (1) — Diarrhoea
Bruising to Left Antecubital Fossa (Venepuncture Related) (General disorders) | 1 (1) — Vessel Puncture Site Bruise
COVID-19 (Infections and infestations) | 1 (1) — COVID-19
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Oropharyngeal Pain
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) — Night Sweats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT06469138/Prot_SAP_000.pdf